CLINICAL TRIAL: NCT03979495
Title: mFOCUS (Multilevel FOllow-up of Cancer Screening)
Acronym: mFOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer S Haas, MD, Peter L. Gross MD Chair in Primary Care, Director of Research and Research Education, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2019P000341
Record Dates: First submitted 2019-05-30; First posted 2019-06-07 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Abnormal Screening Results
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: All individuals in this study will receive the current standard of care at Massachusetts General Hospital, Brigham and Women's Hospital, and Dartmouth Hitchcock for the follow-up of abnormal cancer screening tests (Arms 1-4). In addition to this standard of care, we will test 3 additional arms of increasing intensity of intervention: Arm 2-access to an IT platform to facilitate updates to HM modifiers and problem lists for visit-based reminders; Arm 3- the IT platform in addition to automated reminders to patients between visits and the care team; Arm 4-the IT platform, automated reminders, and administrative outreach and navigation to help with scheduling and to address social barriers to care.
Masking Description: The intervention is not masked to the providers or the participants. Randomization status is masked to the participants but not the providers. Masking is not feasible because randomization will take place at the level of the practice and practices will need to be informed about intervention components that will be made available to patients in their practice and the health care team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of care (No Intervention): standard of care
- IT platform (Active Comparator): Access to an IT platform for visit-based reminders about overdue abnormal cancer screening test results
  Interventions: Other: mFOCUS
- IT platform with reminders (Active Comparator): Access to an IT platform that will deliver both visit based and between visit reminders about abnormal cancer screening test results.
  Interventions: Other: mFOCUS
- IT platform and patient navigation (Active Comparator): the IT platform available in Arm 3 and navigation to help with scheduling and to address social barriers to care.
  Interventions: Other: mFOCUS

INTERVENTIONS:
Other: mFOCUS — To evaluate the effectiveness of the system, team and individual components of mFOCUS vs. standard care by conducting a 4-arm cluster randomized controlled trial (RCT) of individuals who are due for follow-up of an abnormal screen.
  Arms: IT platform; IT platform and patient navigation; IT platform with reminders

SUMMARY:
To evaluate the effectiveness of the system, team and individual components of mFOCUS vs. standard care by conducting a 4-arm cluster randomized controlled trial (RCT) of individuals who are due for follow-up of an abnormal cancer screening test.

DETAILED DESCRIPTION:
Standard care consists of well-characterized existing decision support and systems for follow-up in these three participating primary care networks and their affiliated integrated delivery systems (Brigham and Women's Hospital, Massachusetts General Hospital, and Dartmouth Hitchcock Health, the largest health care provider in New Hampshire). The primary outcome will be whether an individual receives follow-up, defined based on the type of screening abnormality and organ type (breast, cervical, lung or colorectal cancer), within 120 days of becoming eligible for mFOCUS. Secondary comparisons will assess multi- and cross-level (individual, team, system) outcomes. The study design will allow us to examine the marginal effectiveness of system, team and individual-level enhancements, and exploratory analyses will address subgroups defined by race/ ethnicity, socioeconomic status and cancer type.

ELIGIBILITY:
Inclusion Criteria:

individuals who have an abnormal screen that is due for follow-up including:

* Breast: women 40-80 years with an incident (i.e., newly detected) abnormal screening mammogram or digital breast tomosynthesis (DBT) exam.
* Cervical: women 21-65 years with an incident abnormal screening Pap.
* Colorectal: adults 40-80 years with an abnormal screen, including incident FOBT (Fecal Occult Blood Test) / FIT (Fecal Immunochemical Test), or prevalent colonoscopy. Because of the long periods of time required for follow-up of colonoscopies, we will look back over a 5-year period and will therefore find prevalent abnormalities that become due for follow-up.
* Lung: adults 55-80 years, current and former smokers, with an incident abnormal LDCT (Low Dose Computed Topography) result.

Exclusion Criteria:

We will exclude patients who:

* are not English or Spanish-speaking
* have had prior cancer of the organ for each screening test (i.e., women with prior breast cancer will not be tracked for breast cancer screening abnormalities) as these individuals may have non-standard follow-up care recommendations.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11980 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock, Hanover, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atlas SJ, Gallagher KL, McGovern SE, Wint AJ, Smith RE, Aman DG, Zhao W, Burdick TE, Orav EJ, Zhou L, Wright A, Tosteson ANA, Haas JS. Patient Perceptions on the Follow-Up of Abnormal Cancer Screening Test Results. J Gen Intern Med. 2025 May;40(6):1280-1287. doi: 10.1007/s11606-024-09128-4. Epub 2024 Oct 18. PMID 39424768
- [Derived] Atlas SJ, Tosteson ANA, Wright A, Orav EJ, Burdick TE, Zhao W, Hort SJ, Wint AJ, Smith RE, Chang FY, Aman DG, Thillaiyapillai M, Diamond CJ, Zhou L, Haas JS. A Multilevel Primary Care Intervention to Improve Follow-Up of Overdue Abnormal Cancer Screening Test Results: A Cluster Randomized Clinical Trial. JAMA. 2023 Oct 10;330(14):1348-1358. doi: 10.1001/jama.2023.18755. PMID 37815566
- [Derived] Haas JS, Atlas SJ, Wright A, Orav EJ, Aman DG, Breslau ES, Burdick TE, Carpenter E, Chang F, Dang T, Diamond CJ, Feldman S, Harris KA, Hort SJ, Housman ML, Mecker A, Lehman CD, Percac-Lima S, Smith R, Wint AJ, Yang J, Zhou L, Tosteson ANA. Multilevel Follow-up of Cancer Screening (mFOCUS): Protocol for a multilevel intervention to improve the follow-up of abnormal cancer screening test results. Contemp Clin Trials. 2021 Oct;109:106533. doi: 10.1016/j.cct.2021.106533. Epub 2021 Aug 8. PMID 34375748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in August 2020 and ended in December of 2021
Units Other Than Participants: Primary Care Practices
Groups:
- Standard of Care: Standard care/no changes to usual care
Period: Overall Study
Arm/Group | Standard of Care | IT Platform | IT Platform With Reminders | IT Platform and Patient Navigation
Started | 2702; 11 Primary Care Practices | 3254; 11 Primary Care Practices | 2569; 11 Primary Care Practices | 3455; 11 Primary Care Practices
Completed | 2702; 11 Primary Care Practices | 3254; 11 Primary Care Practices | 2569; 11 Primary Care Practices | 3455; 11 Primary Care Practices
Not Completed | 0; 0 Primary Care Practices | 0; 0 Primary Care Practices | 0; 0 Primary Care Practices | 0; 0 Primary Care Practices

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | IT Platform | IT Platform With Reminders | IT Platform and Patient Navigation | Total
Number analyzed (Participants) | 2702 | 3254 | 2569 | 3455 | 11980
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1828 | 2051 | 1557 | 2042 | 7478
  >=65 years | 874 | 1203 | 1012 | 1413 | 4502
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1772 | 2139 | 1680 | 2172 | 7763
  Male | 930 | 1115 | 889 | 1283 | 4217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 207 | 316 | 228 | 344 | 1095
  Not Hispanic or Latino | 2310 | 2642 | 2137 | 2913 | 10002
  Unknown or Not Reported | 185 | 296 | 204 | 198 | 883
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 7 | 6 | 12 | 29
  Asian | 90 | 89 | 77 | 101 | 357
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 2 | 6
  Black or African American | 139 | 265 | 184 | 201 | 789
  White | 2241 | 2546 | 2051 | 2782 | 9620
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 226 | 346 | 250 | 357 | 1179
Region of Enrollment [Number; unit: participants]
  United States | 2702 | 3254 | 2569 | 3455 | 11980

OUTCOME MEASURES:

1. Primary Outcome: Completion of Follow-up Test
Description: Completion of follow-up test within 120 days of eligibility for mFOCUS (EHR)
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | IT Platform | IT Platform With Reminders | IT Platform and Patient Navigation
Number analyzed (Participants) | 2702 | 3254 | 2569 | 3455
Participants | 672 | 796 | 831 | 1062

2. Secondary Outcome: Number of Participants Who Complete the Required Diagnostic Evaluation
Description: How many participants completed the required diagnostic evaluation (EHR), 0-60, 61-120, 121-180, 181-240 day intervals were evaluated.
Time Frame: up to 240 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | IT Platform | IT Platform With Reminders | IT Platform and Patient Navigation
Number analyzed (Participants) | 2702 | 3254 | 2569 | 3455
Participants
  0-60 days | 423 | 464 | 514 | 653
  61-120 days | 249 | 332 | 317 | 409
  121-180 days | 170 | 215 | 191 | 255
  181-240 days | 113 | 159 | 100 | 153
  Did not receive follow up | 1747 | 2084 | 1447 | 1985

ADVERSE EVENTS:
Time Frame: 240 days
Arm/Group | Standard of Care | IT Platform | IT Platform With Reminders | IT Platform and Patient Navigation
All-Cause Mortality (participants affected / at risk) | 0/2702 | 0/3254 | 0/2569 | 0/3455
Serious Adverse Events (participants affected / at risk) | 0/2702 | 0/3254 | 0/2569 | 0/3455
Other Adverse Events (participants affected / at risk) | 0/2702 | 0/3254 | 0/2569 | 0/3455

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT03979495/Prot_SAP_000.pdf